CLINICAL TRIAL: NCT05109156
Title: Preoperative Sepsis Timeline, Profile and Its Association With Recipient Outcome Following Live Donor Liver Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Sepsis-02
Record Dates: First submitted 2021-10-20; First posted 2021-11-05 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-10

CONDITIONS: Sepsis; Liver Transplant; Complications
Keywords: Sepsis; Live donor liver transplant(LDLT),; Liver capsular macrophages(LCM); Peritoneal macrophages(PM)
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Explant liver with be sent for assessment of the subcapsular layer in addition to routine Histo pathological examination (HPE).
  20 ml of peritoneal fluid from the recipient will also be collected and processed for analysis of peritoneal macrophages.
  Samples will then be subjected to flow cytometry for assessment of:
  1. Macrophage identification markers: Quantitative assessment .
  2. Macrophage Activation markers: Qualitative/ Activation assessment. Density and functionality of both LCM and PM will then be co-related to both pre-LT sepsis timeline and profile as well as post operative recipient outcome .
  Identification of Macrophage populations using Flow Cytometry and Immunohistochemistry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This is an observational study: This is an observational study
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study — This is an observational study

SUMMARY:
Preoperative sepsis timeline, profile and its association with recipient outcome following live donor liver transplant.

DETAILED DESCRIPTION:
Sepsis is a critical factor causing major mortality and morbidity in liver recipients.

* According to guidelines patients with active infection should be treated before listing, and those who develop infection while on the waiting list should be removed until the infection is cured or has improved with appropriate antimicrobial treatment.
* Live donor liver transplant (LDLT) in comparison to Deceased Donor Liver Transplant (DDLT) is a more planned surgery. This gives us an opportunity for preoperative optimization and surgery can be timed. In identifying the impact of timing of LDLT wrt. sepsis , major morbidity can be reduced by optimizing/delaying timing of transplant. On the other hand, preoperative optimization may not be as critical as currently thought, and many more patients , currently delisted following sepsis can reap the benefits of a timely transplant. Results will help in better selection of patients as well as better management of pre transplant sepsis. A variety of studies have evaluated the impact of preoperative sepsis at different periods prior to LT on postoperative outcomes but results are widely varied.

The subsets of macrophages in hepatic capsule are known as liver capsular macrophages(LCMs). LCMs recruit neutrophils in response to bacteria reaching the liver capsule .LCM depletion increases liver pathogen load. Further it is also important to study peritoneal macrophages in chronic liver disease . Chronic sterile inflammation, as in nonalcoholic fatty liver disease, is associated with constant release of damage-associated molecular patterns. Continuous activation and recruitment of peritoneal and Liver capsular macrophages may contribute to fibrogenesis under condition of chronic liver diseases. Study of LCMs and PMs could be a landmark study identifying peritoneal macrophages and Liver capsular macrophages as highly mobile cells with a specialized function , with many possible therapeutic applications.The study will be collecting data both prospectively and retrospectively and will involve assessment of association of timeline and profile of preoperative sepsis on mortality and morbidity of liver transplant recipients. Primary objective will be Correlation of timeline of sepsis with recipient outcome following Live donor liver transplant. Outcome parameters will be Post operative sepsis ,In hospital mortality, Hospital stay, ICU stay, Retransfer to ICU, Days on ventilator, Need for tracheostomy/re-intubation, Duration of inotropic support. Secondary objectives To study the impact of source of sepsis on postoperative outcomes, To evaluate the causative organism of sepsis on post operative outcome. To study the correlation between recipient liver capsular and peritoneal macrophage activity and preoperative sepsis timeline, profile as well as post operative recipient outcome. 25 samples will be collected for liver capsular and peritoneal macrophage study.

ELIGIBILITY:
Inclusion Criteria:All patients who undergo living donor liver transplant.

-

Exclusion Criteria: Acute Liver Failure

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing/ undergone live donor liver transplant at our institute
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of timeline of sepsis with recipient outcome following Live donor liver transplant. | 30 days
  a. Post-operative sepsis b. In hospital mortality c. Hospital stay d. ICU stay e. Retransfer to ICU f. Days on ventilator g. Need for tracheostomy/re-intubation h Duration of inotropic support

SECONDARY OUTCOMES:
study the correlation between recipient liver capsular and peritoneal macrophage activity and preoperative sepsis timeline, profile as well as post operative recipient outcome. | 30 days
  study the correlation between recipient liver capsular and peritoneal macrophage activity and preoperative sepsis timeline, profile as well as post operative recipient outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, FEBS, Study Director — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided